CLINICAL TRIAL: NCT03857763
Title: A Prospective Study of Apatinib Plus Concurrent Neoadjuvant Chemoradiotherapy in Patients With Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBAE-01
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib+Paclitaxel+Cisplatin+RT (Experimental): Apatinib：250mg,po,qd, d1-35; Paclitaxel：50mg/m2 iv, d1，8，15，22，29; Cisplatin: 30mg/m2 iv, d1，8，15，22，29; Radiotherapy：41.4Gy/23f , 1.8Gy/f，5 f/w
  Interventions: Combination Product: Apatinib,Paclitaxel,Cisplatin,RT

INTERVENTIONS:
Combination Product: Apatinib,Paclitaxel,Cisplatin,RT — Apatinib Mesylate Tablets 250mg qd p.o. d1-35; Paclitaxel：50mg/m2 iv d1，8，15，22，29; Cisplatin: 30mg/m2 iv d1，8，15，22，29; RT：41.4Gy/23f , 1.8Gy/f，5 f/w

SUMMARY:
The purpose of this study is to assess the efficacy and safety of apatinib plus concurrent neoadjuvant chemoradiotherapy in patients with esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 70 years old (man or female);
2. Pathologically diagnosed with esophageal squamous cell carcinoma;
3. Patients with Stage for Ⅱ-Ⅲ(T2-4N0/+M0) (According to transesophageal ultrasonography;
4. Patients with measurable lesions(According to the criteria in RECIST1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
6. Life expectancy greater than or equal to 3 months;
7. Major organ function has to meet the following certeria:

(1) For results of blood routine test

1. HB≥80g/L;
2. ANC≥1.5×109/L;
3. PLT≥90×109/L; (2) For results of blood biochemical test

a) ALT and AST≤2.5×ULN; b) TBIL<1.5×ULN; c) Serum creatinine ≤1.5×ULN; 8. Doctors believe that treatment can bring benefits to patients; 9. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Have received prior treatment with chemotherapy or radiotherapy；
2. Have high blood pressure and antihypertensive drug treatment can not control;
3. Patients with severe cardiovascular disease ;
4. Accompanied by esophageal perforation and esophagotracheal fistula;
5. Patients with active bleeding or bleeding tendency;
6. Pregnant or lactating women;
7. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response rate(pCR) | within 3 weeks after surgery
  The lesion disappeared completely by pathology

SECONDARY OUTCOMES:
R0-resection rate | within 3 weeks after surgery
  There was no residual by the microscope
Disease-free survival(DFS) | 3 years
  Baseline to measured date of recurrence or death from any cause
Overall survival (OS) | 1year
  Baseline to measured date of death from any cause
Adverse events Toxicity | 3 years
  Adverse events Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.The number of Participants with adverse events will be recorded at each treatment visit.

IPD SHARING:
Plan to Share IPD: No